CLINICAL TRIAL: NCT06663306
Title: Efficacy and Safety of Pemetrexed Combined With Bevacizumab Intrathecal Injection in Patients With Leptomeningeal Metastases in NSCLC
Brief Title: Intrathecal Injection Pemetrexed And Bevacizumab in Patients With Leptomeningeal Metastases in NSCLC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Hua Zhong, Chief of Respiratory Department, Shanghai Chest Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS24103
Record Dates: First submitted 2024-10-24; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer (NSCLC); Leptomeningeal Metastasis
Keywords: Leptomeningeal Metastases; NSCLC; Intrathecal Injection
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Meningeal Carcinomatosis | interventions — Pemetrexed; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Enrolled patients were treated with pemetrexed intrathecal injection
  Interventions: Drug: Pemetrexed
- Arm B (Experimental): Enrolled patients were treated with pemetrexed combined with bevacizumab intrathecal injection
  Interventions: Drug: Pemetrexed; Drug: Bevacizumab

INTERVENTIONS:
Drug: Pemetrexed — Intrathecal pemetrexed 50mg,twice per week (d1, d8) for 1 week, then once per 4 weeks
Drug: Bevacizumab — Intrathecal bevacizumab, once (d8)for 1 week, then once per 4 weeks.The initial dose of intrathecal bevacizumab is 5 mg, escalated to 10 mg, and then 25 mg, and then 37.5mg, and then 50mg.
  Arms: Arm B

SUMMARY:
This is a prospective, single-arm, phase Ia clinical study, which was designed to evaluate the efficacy and safety of Pemetrexed Combined With Bevacizumab Intrathecal Injection in Patients With Leptomeningeal Metastases in NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* ECOG PS score 0-3. ECOG PS score 2 or 3 should be due to leptomeningeal metastases.
* Patients with pathologically diagnosed non-small cell lung cancer with cerebrospinal fluid and/or MRI diagnosis of leptomeningeal metastasis(LM);
* Unsatisfactory efficacy of LM,which defined as disease progression in LM,or LM-related neurological progression, while patients received standard systemic anti-tumor treatment;
* Expected survival time ≥ 1 month;
* The laboratory test results meet the following criteria:Hemoglobin ≥ 90 g/L, neutrophil count ≥ 1.5 × 10^9/L, platelet count ≥ 100 × 10^9/L; Total bilirubin ≤ 1.5 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN ; Creatinine≤ 2.0 × ULN,or Creatinine clearance rate (CrCl) ≥ 50 mL/min;
* Females of child-bearing potential agree to use contraception during the study period and for 6 months after the completion of the study; patients who have had a negative serum or urine pregnancy test within seven days prior to enrollment in the study and who are not breastfeeding; and males agreeing to use contraception during the study period and for 6 months after the completion of the study;
* Understand and sign the informed consent form.

Exclusion Criteria:

* Positive for human immunodeficiency virus (HIV) ;
* History of allergy to pemetrexed or bevacizumab;
* History of pemetrexed and/or bevacizumab intrathecal Injection;
* Presence of contraindication of bevacizumab:

  1. Uncontrolled hypertension(systolic pressure≥150mmHg，or diastolic pressure≥100mmHg；History of hypertensive crisis or hypertensive encephalopathy;
  2. Urine protein≥2+,or 24-hour urine protein≥2g；
  3. Unstable angina pectoris, symptomatic congestive heart failure,myocardial infarction within 6 months before enrollment, severe vascular disease, severe uncontrolled arrhythmia;
  4. Major hemoptysis within the past 1 month; History of coagulation disorders;
  5. Presence of serious non-healing wounds, ulcers, or bone fractures
  6. Presence of abdominal fistula, gastrointestinal perforation, or gastrointestinal tract obstruction;
  7. Presence of macrovascular invasion；
  8. Some neurological disorders unrelated to tumors，such as intracranial infection,cerebral hemorrhage,cerebral infarction,encephalitis;
* Brain/spinal cord radiation therapy within 1 week before enrollment;
* Pregnant and lactating female;
* Refuse to use contraception during the study period;
* Individuals considered by the investigator to be unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (Safety and Tolerability) | From the beginning of the treatment until two months after the treatment.
  Number of participants with adverse events, treatment emergent adverse events,and serious adverse events assessed by CTCAE v5.0 as a measure of safety and tolerability.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 2 years
  Kaplan-Meier method used to estimate the distribution of OS from the start of study treatment.

OTHER OUTCOMES:
Clinical response rate | Up to 2 years
  The evaluation of clinical response rate was assessed by the investigators, which based on improvement of neurologic symptoms/signs and changes in the Karnofsky performance status score . This evaluation consists of five layers, including complete response (CR), obvious response (OR), partial response (PR), stable disease (SD) and progressive disease (PD).Clinical response was defined as the continuous presence of CR, OR or PR within an interval of at least 1 week. SD and PD were defined as ineffective.
CSF cytology | From the beginning of the intrathecal treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  Cerebrospinal fluid (CSF) was collected before each cycle of intrathecal treatment, and assessed by the investigators the presence of tumor cells (Positive or Nagetive).
Radiographic assessment | From the beginning of the treatment until two months after the treatment.
  Radiographic assessment with complete contrast-enhanced neuro-axis MRI or CT, Leptomeningeal metastases response was evaluated using the Response Assessment in Neuro-Oncology (RANO) criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China